CLINICAL TRIAL: NCT01642641
Title: The Efficacy of Different Surgical Modalities in the Treatment of Periodontitis. A Randomised Controlled Trial
Brief Title: Different Surgical Modalities in the Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 011467; COCR0003 (Other: QMUL)
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-surgical subgingival debridement (Active Comparator)
  Interventions: Procedure: Non-surgical Subgingival Debridement (SD)
- Simplified Papilla Preservation Flap (Active Comparator)
  Interventions: Procedure: Simplified Papilla Preservation Flap
- Resective Flap with Osseous Recontouring (Active Comparator)
  Interventions: Procedure: Resective Periodontal Flap with Osseous Recontouring (RPFO)

INTERVENTIONS:
Procedure: Non-surgical Subgingival Debridement (SD) — SD is a conservative non-surgical procedure aimed at reducing dental plaque and calculus from the tooth root usually under local anaesthesia.
  Arms: Non-surgical subgingival debridement
Procedure: Simplified Papilla Preservation Flap — The simplified papilla preservation flap is a novel conservative surgical procedure aimed at the preservation of the tissues between the teeth. It has been shown to significantly reduce pocket depth and has faster re-vascularisation of the flap, when compared with other procedures.
  Arms: Simplified Papilla Preservation Flap
Procedure: Resective Periodontal Flap with Osseous Recontouring (RPFO) — RPFO is a surgical procedure that involves the resection of soft and hard tissue to obtain optimum tissue architecture and pocket reduction or elimination.
  Arms: Resective Flap with Osseous Recontouring

SUMMARY:
The purpose of the present study is to determine: 1) the efficacy of 2 periodontal surgical procedures, the conservative simplified papilla preservation technique and the more resective open flap debridement with osseous recontouring, in the treatment of chronic periodontitis in terms of clinical, radiographic, microbiological, immunological and PROMs, comparing them to non-surgical subgingival debridement and 2) if possible, determine the surgical procedure which leads to pocket elimination or to the lowest number of residual pockets.

DETAILED DESCRIPTION:
Periodontal diseases (PD) are highly prevalent chronic diseases, and may be associated with loss of gum and bone tissue surrounding the tooth. Among adults (with 2 or more teeth remaining) in England, 54% experienced gum bleeding and 45% had periodontal (gum) disease of which 9% was severe. Bacterial in origin, the high prevalence of PD, together with increased retention of teeth at older ages, has considerable implications for the population's future treatment needs and the associated costs to the health system. It is therefore important to ensure interventions delivered are those proven to be most efficient and cost effective. The investigators study question will therefore be, "In an adult population with moderate to severe chronic periodontitis, how will 3 different treatment approaches; simplified papilla preservation flap (SPPF), resective periodontal flap with osseous recontouring (RPFO) and subgingival debridement (SD), differ in regard to healing and resolution of disease, patient reported outcomes and cost effectiveness?" The aim of this study is to find the most efficient way to treat chronic periodontitis, through a multi-centre randomised, single-blind, parallel- surgical modalities groups (3 groups) clinical trial including 3 sites:: 1. QMUL Institute of Dentistry, Centre for Oral Clinical Research (COCR) as the new sponsor and coordinating centre including overarching custodian responsibilities for samples and data collected. 2. Barts Health NHS Trust Dental Hospital where the trial different surgical modalities will take place going forward for all new patients recruited. 3. UCL Eastman Dental Institute where patients already recruited and completed the trial surgical phase will complete their follow up.

A sufficient number of adults (29 per group) presenting; a total of 87 patients with chronic periodontitis and meeting the necessary inclusion and exclusion criteria will be entered into the trial. Subjects will present to the clinical site for initial screening and enrolment (Baseline Visit). Following enrolment, all participants will attend one visit as preparation for the subsequent study treatments. As part of this session, participants will review how to perform efficient self-care regimes at home to remove plaque biofilm accumulations on a regular basis. At this appointment, they will be randomised to their assigned treatment group and the pending treatment will be discussed with them. Treatment groups will consist of simplified papilla preservation flap (SPPF), resective periodontal flap surgery with osseous recontouring (RPFO), or non-surgical subgingival debridement with local anaesthesia (SD). Treatment will take place within 4 weeks of this preparation visit. Participants will then attend for follow-up visits at 1, 2, 3 and 4 weeks post treatment for evaluation of healing, reinforcement of oral hygiene regime, and supra-gingival scale and polish as required. Clinical measurements will be recorded again at 3, 6 and 12 months post treatment. Radiographs will be taken at baseline, and 12 months post treatment. A saliva and plaque sample will be taken at baseline, 3, 6 and 12 months post treatment. GCF will be taken at baseline, 2 weeks and 3 months post treatment. Patient reported outcomes will be evaluated at baseline, 1 week, 3, 6, 9 and 12 months post treatment. Use of NHS and private dental and health services will be collected via self-reported patient diaries distributed at the first intervention appointment, and 3, 6 and 9 months post intervention. Supportive periodontal maintenance visits will be carried out every 3 months for the duration of the study to maintain optimal oral health through monitoring of oral hygiene routine and supra and subgingival scaling and polish as required. A dental prophylaxis will be performed at the end of the study and the study termination form will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy males and females ≥ 30 years of age.
2. Volunteers must be willing to read, and sign a copy of the Informed Consent Form after reading the Patient Information Leaflet and after the nature of the study has been fully explained.
3. Present with clinical evidence of periodontitis, with one interdental area of PPD ≥6mm, BOP, and attachment loss ≥6mm in any posterior sextant of their mouth (excluding third molars and distal of second molars), or multiple sites (≥9) with PPD ≥5mm, BOP, and attachment loss ≥5mm.
4. Have completed a course of non-surgical periodontal therapy within 2 years prior to study commencement and have had maintenance subgingival debridement within 6 months prior to assessment for eligibility.

Exclusion Criteria:

1. Medical history that includes diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases e.g. cardiovascular disease or AIDS.
2. History of rheumatic fever, heart murmur, mitral valve prolapse, artificial heart valve or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
3. Antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam.
4. History of alcohol or drug abuse.
5. Self reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).
6. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of 3 different periodontal treatment approaches | 3, 6 and 12 months
  A clinical measure of resolution of disease from baseline in Periodontal Probing Depths (PPD)
Change from Baseline of EuroQol-5D-5L and Condition Specific Oral Impacts on Daily Performance Questionnaire | Baseline, 1 week post-op, 3, 6, 9 and 12 months
  To assess impact on quality of life.

SECONDARY OUTCOMES:
To investigate the efficacy of 3 different periodontal treatment approaches on PROMs related to general health over a follow-up period of 12 months | Treatment Visit 1, 3, 6 and 9 months
  To assess impact on general health
Incremental cost per quality-adjusted life year gained | 3, 6, 9 and 12 months
  To determine cost-effectiveness from an NHS perspective
Maintenance/support needs of patients following treatment | 3, 6 and 12 months
  Measurement of effectiveness of study different treatments
Radiographic bone changes of 3 different periodontal treatment approaches | Baseline and 12 months
  Linear measurements obtained from standardized peri-apical radiographs
Changes in subgingival microbiota | Baseline, 3, 6 and 12 months
  Assessed via pooled samples and analyzed via Illumina Miseq sequencer
To investigate changes from baseline in saliva inflammatory biomarkers and protein expression | Baseline, 3, 6 and 12 months
  Proteomic analysis of saliva with LC/MS (liquid chromatography/tandem mass spectrometry)
Facial changes in post-operative swelling and oedema | Right before treatment, 1 week and 2 weeks post-operatively
  Measurement with 3D imaging technique at different time points following the different periodontal treatments
To identify the preferred intervention for subgroups of patients based on severity of disease at presentation to secondary care | Treatment Visit 1, 3, 6 and 9 months
  Assess patient's preference of treatment modality
To explore whether outcomes measured at 3 months are sufficiently robust predictors of long-term outcome to be useful in patient management and for monitoring in a timely manner the outcomes being achieved in secondary care | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, DDS, MS, PhD, Study Director — Barts & The London School of Medicine & Dentistry, QMUL; Nikolaos Mardas, DDS, MS, PhD, Principal Investigator — Barts & The London School of Medicine & Dentistry, QMUL; Natalie M Leow, BDS, MDSc, Principal Investigator — UCL Eastman Dental Institute
Locations (3):
- United Kingdom (3):
  - Barts Health NHS Trust Dental Hospital, London
  - Centre for Oral Clinical Research, London
  - Eastman Clinical Investigation Centre, London